CLINICAL TRIAL: NCT02204891
Title: A Clinical Study of the Efficacy of a Formulation of Four Probiotics in Patients With Syndrome of Intestinal Bacterial Overgrowth and Irritable Bowel Syndrome
Brief Title: Probiotics in Intestinal Bacterial Overgrowth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Evangelos J. Giamarellos-Bourboulis, M.D., Associate Professor of Medicine, University of Athens
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LACTO01
Record Dates: First submitted 2014-07-28; First posted 2014-07-31 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: Abdominal pain; Abdominal discomfort; Flatulence; Diarrhea; Bacterial overgrowth; Cytokines
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain; Flatulence; Diarrhea | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics in SIBO (Experimental): Administration of probiotics in patients with IBS and SIBO
  Interventions: Dietary Supplement: Probiotics in SIBO
- Probiotics (Active Comparator): Administration of probiotics in patients with IBS without SIBO
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics in SIBO — Mixture of the four probiotics in one capsule. One capsule twice daily for 30 days
  Other Names: Saccharomyces Bifidobacterium Lactobacillus species
  Arms: Probiotics in SIBO
Dietary Supplement: Probiotics — One capsule twice daily for 30 days
  Arms: Probiotics

SUMMARY:
The aim of the present study is to demonstrate the effect of a mixture of four species of probiotics (Saccharomyces boulardii, Bifidobacterium lactis BB-12, Lactobacillus acidophilus LA-5 and Lactobacillus plantarum) in patients with symptomatic irritable bowel syndrome (IBS) who have culture verified syndrome of intestinal bacterial overgrowth (SIBO) and those who do not have. This will provide direct evidence for the role of probiotics in treating part of the pathogenesis of IBS.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is the most common gastrointestinal disorder. Pathogenesis remains multifactorial. Better understanding of the interaction of the host with intestinal microbiota the last decade led to the knowledge that many of the symptoms of IBS, mainly bloating and diarrhea, are related with the overgrowth of bacteria of colonic type in the small intestine. This overgrowth frames the syndrome of intestinal bacterial overgrowth (SIBO) where colonic type of bacteria predominate in the proximal parts of the small intestine. Fermentation of dietary carbohydrates by the bacteria colonizers of SIBO ends with the over-production of gas generating thus symptoms of IBS. The relationship between IBS and SIBO was found by a series of prospective observational studies using the lactulose and the glucose tolerance tests for the diagnosis of SIBO. Using this test, the prevalence of SIBO in patients with IBS ranged between 65 and 85%. The gold-standard technique for the diagnosis of SIBO is the quantitative culture of the content of the proximal intestine i.e. of the duodenum after upper GI tract endoscopy. Few studies are available with this design and they suggest a growth of colonic type of flora at counts equal to or greater than 10^5 cfu/ml as diagnostic of SIBO. Based on systematic review of the literature but also on data generated in a cohort of 320 consecutive patients undergoing upper GI tract endoscopy, normal subjects are never greater than 10^3 cfu/m in the duodenum. In the latter publication coming from Athens, using variable cut-offs greater than 10^3 or 10^4 or 10^5 cfu/ml for the diagnosis of SIBO, the frequency of SIBO was significantly greater among sufferers than among non-sufferers from IBS.

Oral supplementation with probiotics may be a rational approach for the eradication of SIBO and subsequently of the symptoms of IBS. The majority of probiotic bacteria belong to the Lactobacillus and Bifidobacterium genera. They are Gram-positive lactic acid-producing bacteria that constitute a major part of the normal intestinal microflora in animals and humans. The rationale behind their use as a therapeutic strategy in IBS is that orally administered probiotics may replace the overgrown enteric-type bacteria of SIBO. Four randomized clinical trials are available evaluating the efficacy of orally administered probiotics in IBS. The common findings of these trials are that a) efficacy refers to the improvement of symptoms of bloating and of diarrhea that are typical symptoms of the presence of SIBO; and b) efficacy is usually found when mixtures of different species of probiotics are used. However, no study has ever tested the efficacy of probiotics in patients with IBS and SIBO proven by small intestinal culture.

The aim of the present study is to demonstrate the effect of a mixture of four species of probiotics (Saccharomyces boulardii, Bifidobacterium lactis BB-12, Lactobacillus acidophilus LA-5 and Lactobacillus plantarum) in patients with symptomatic IBS who have culture verified SIBO and those who do not have. This will provide direct evidence for the role of probiotics in treating part of the pathogenesis of IBS.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Both genders
3. Written informed consent by study participants
4. Presence of IBS according to Rome III criteria
5. Equal number of SIBO-positive and SIBO-negative patients

Exclusion Criteria:

1. Age <18 years
2. Deny to consent
3. Pregnancy or lactation
4. Presence of inflammatory bowel disease
5. Presence of acute GI tract infection
6. Diabetes mellitus type 1 or type 2
7. Use of laxatives and antibiotics within the preceding 6 weeks
8. Presence of fever, abdominal mass, signs of bowel obstruction and/or leucocytosis
9. Abnormal serum levels of thyroid -stimulating hormone.
10. History of colon cancer or diverticulitis
11. Infection by human immunodeficiency virus (HIV), hepatitis B virus and hepatitis C virus
12. Patients with celiac disease defined by biopsy of the duodenal mucosa.
13. History of scleroderma and gastroparesis
14. Pregnancy or planning pregnancy the next 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
• The efficacy of probiotics in improvement of symptoms of IBS in patients with SIBO compared to their efficacy in patients with IBS without SIBO. | 30 days
  This will be assessed after 30 days from start of therapy (visit 2) by comparisons of grading of symptoms and results of OLT between the two groups of treatment.

SECONDARY OUTCOMES:
• The efficacy of probiotics in symptoms of IBS in patients with SIBO compared to their efficacy in patients with IBS without SIBO. | 60 days
  This will be assessed after 60 days from start of therapy (visit 3) by comparisons of grading of symptoms and results of OLT between the two groups of treatment.
The efficacy of probiotics in specific symptoms of IBS both visits 2 and 3. | Days 30 and 60
  This will be done by comparing the grading for every symptom of IBS of patients in visits 2 and 3 compared with the baseline visit 1.
• The importance of the inflammation cascade in the pathogenesis of SIBO-related IBS. | 30 days
  This will be done by comparing the duodenal aspirate cytokines of the two groups of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Triantafyllou, MD, PhD, Principal Investigator — University of Athens, Medical School; Evangelos Giamarellos-Bourboulis, MD, PhD, Principal Investigator — University of Athens, Medical School
Locations (1):
- Department of Gastroenterology, ATTIKON University Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pyleris E, Giamarellos-Bourboulis EJ, Tzivras D, Koussoulas V, Barbatzas C, Pimentel M. The prevalence of overgrowth by aerobic bacteria in the small intestine by small bowel culture: relationship with irritable bowel syndrome. Dig Dis Sci. 2012 May;57(5):1321-9. doi: 10.1007/s10620-012-2033-7. Epub 2012 Jan 20. PMID 22262197
- [Background] Choi CH, Jo SY, Park HJ, Chang SK, Byeon JS, Myung SJ. A randomized, double-blind, placebo-controlled multicenter trial of saccharomyces boulardii in irritable bowel syndrome: effect on quality of life. J Clin Gastroenterol. 2011 Sep;45(8):679-83. doi: 10.1097/MCG.0b013e318204593e. PMID 21301358
- [Background] Ringel-Kulka T, Palsson OS, Maier D, Carroll I, Galanko JA, Leyer G, Ringel Y. Probiotic bacteria Lactobacillus acidophilus NCFM and Bifidobacterium lactis Bi-07 versus placebo for the symptoms of bloating in patients with functional bowel disorders: a double-blind study. J Clin Gastroenterol. 2011 Jul;45(6):518-25. doi: 10.1097/MCG.0b013e31820ca4d6. PMID 21436726
- [Background] Ki Cha B, Mun Jung S, Hwan Choi C, Song ID, Woong Lee H, Joon Kim H, Hyuk J, Kyung Chang S, Kim K, Chung WS, Seo JG. The effect of a multispecies probiotic mixture on the symptoms and fecal microbiota in diarrhea-dominant irritable bowel syndrome: a randomized, double-blind, placebo-controlled trial. J Clin Gastroenterol. 2012 Mar;46(3):220-7. doi: 10.1097/MCG.0b013e31823712b1. PMID 22157240
- [Background] Yoon JS, Sohn W, Lee OY, Lee SP, Lee KN, Jun DW, Lee HL, Yoon BC, Choi HS, Chung WS, Seo JG. Effect of multispecies probiotics on irritable bowel syndrome: a randomized, double-blind, placebo-controlled trial. J Gastroenterol Hepatol. 2014 Jan;29(1):52-9. doi: 10.1111/jgh.12322. PMID 23829297
- [Derived] Leventogiannis K, Gkolfakis P, Spithakis G, Tsatali A, Pistiki A, Sioulas A, Giamarellos-Bourboulis EJ, Triantafyllou K. Effect of a Preparation of Four Probiotics on Symptoms of Patients with Irritable Bowel Syndrome: Association with Intestinal Bacterial Overgrowth. Probiotics Antimicrob Proteins. 2019 Jun;11(2):627-634. doi: 10.1007/s12602-018-9401-3. PMID 29508268